CLINICAL TRIAL: NCT04115306
Title: Ph 1/1b/2 Multicenter, Open-Label, FIH Dose Esc & Dose Exp Study to Assess Safety and Tolerability of Orally Administered PMD-026 as a Single Agent and in Combination in Patients With Metastatic or Locally Advanced (Inoperable) RSK2+ Breast Cancer
Brief Title: Phase 1/1b/2 Study of Oral PMD-026 in Patients With Metastatic Breast Cancer
Acronym: Dauntless-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Phoenix Molecular Designs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMD-026-1-001
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer
Keywords: invasive breast cancer; PR-negative breast cancer; HER2-negative breast cancer; Breast cancer; Breast malignancy; breast malignancies; metastatic breast cancer; advanced breast cancer; solid tumor; late stage breast cancer/late-stage breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral PMD-026 in combination with fulvestrant (Experimental): Daily dosing of PMD-026 with fulvestrant dosing according to package insert
  Interventions: Drug: PMD-026; Drug: fulvestrant

INTERVENTIONS:
Drug: PMD-026 — Investigational Drug
Drug: fulvestrant — SERDs
  Other Names: Faslodex

SUMMARY:
The purpose of this study is to test the safety and tolerability of PMD-026 in patients with metastatic breast cancer. PMD-026 is a targeted oral agent designed to kill tumor cells in metastatic breast cancer.

DETAILED DESCRIPTION:
Combination with fulvestrant (Part 3):

This study will enroll RSK2+, HR+, and human epidermal growth factor receptor 2 negative (HER2-) patients to evaluate PMD-026 in combination with a standard dose and schedule of fulvestrant. Fulvestrant will be dosed per the package insert in combination with PMD-026 at the RP2D determined in the monotherapy phase of the study. Up to 20 patients will be enrolled with locally advanced or metastatic HR+/HER2- breast cancer previously treated with a CDK4/6 inhibitor in combination with endocrine therapy.

ELIGIBILITY:
Inclusion Criteria, Combination with fulvestrant (Part 3):

* RSK2 positive from available archival or fresh tumor tissue (FFPE).
* Histologically or cytologically diagnosed HR+, HER2-
* ESR1 wild type
* Diagnosis of adenocarcinoma of the breast with evidence of either locally advanced disease not amendable to resection or radiation with curative intent or metastatic disease not amendable to curative therapy
* Must be appropriate candidates for endocrine therapy
* Previously received at least 1 line of endocrine therapy for MBC or had recurrence while on adjuvant endocrine therapy for locally advanced breast cancer
* Discontinued endocrine therapy at least 15 days prior to first dose of PMD-026
* At least 1 measurable target lesion as defined by RECIST v1.1
* Progression on or after treatment with a CDK4/6 inhibitor in combination with endocrine therapy inhibitor in the locally advanced or metastatic setting
* Adequate hematologic, hepatic, and renal function as assessed by laboratory parameters
* Toxicity related to prior therapy resolved to at least Grade 1 (alopecia excepted) or to at least Grade 2 with prior approval of the Medical Monitor

Exclusion Criteria, Combination with fulvestrant (Part 3):

* Prior chemotherapy
* ESR1 mutations
* ≤14 days from biological or investigational therapy
* Presence of visceral crisis or uncontrolled visceral disease for which chemotherapy would be indicated
* Central nervous system metastases, unless appropriately treated and neurologically stable
* History of leptomeningeal metastases
* Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* Known hepatitis B or hepatitis C infection
* Known HIV-positive with CD4+ cell counts <350 cells/μL
* Known HIV-positive with a history of an AIDS-defining opportunistic infection
* History of clinically significant cardiovascular abnormalities, including QTcF interval >460 msec (using Fridericia's formula)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of PMD-026 in combination with fulvestrant in patients with HR+/HER2- previously treated breast cancer | 6 weeks
  Incidence of AEs, DLTs, SAEs. Changes in laboratory, vital signs, and ECG values.

SECONDARY OUTCOMES:
Plasma concentration of PMD-026 when administered in combination with fulvestrant | As determined by PK data
  The plasma concentration will be measured as part of pharmacokinetic (PK) testing.
Preliminary anti-tumor activity of PMD-026 when dosed in combination with fulvestrant | Until PD or death, up to 2 years
  ORR, DOR, DCR, PFS

OTHER OUTCOMES:
Assess OS | Throughout study
  OS defined as time from first dose to death
Evaluate QT interval and PMD-026 concentrations | Throughout study
  Qualitative and/or quantitative associations of PK parameter concentrations with QTcF changes

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - City of Hope Orange County, Lennar, Irvine, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - City of Hope Chicago, Zion, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Profound Research, Farmington Hills, Michigan
  - Ohio State University, Columbus, Ohio
  - Oncology Consultants, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No